CLINICAL TRIAL: NCT05984680
Title: User-Centered Design of a COPD Care Pathway for Patients With Cancer
Brief Title: COPD Care Pathway Among Patients With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00120161; P30CA012197 (NIH); ONC-LUN-2406 (Other: Wake Forest Baptist Comprehensive Cancer Center); K12TR004931 (NIH)
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Cancer; Head and Neck Cancer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Observational Phase 1: Participants complete surveys
  Interventions: Other: Observational Phase 1
- Observational Phase 2, Group I: Participants complete an interview and participate in a focus group on study.
  Interventions: Other: Observational Phase 2, Group I
- Observational Phase 2, Group II: Participants complete an interview and participate in guided tours of the oncology clinic on study.
  Interventions: Other: Observational Phase 2, Group II
- Observational Phase 3: A subset of interested participants from Phase 2 participate in a workshop on study to develop a final draft of the COPD care pathway.
  Interventions: Other: Observational Phase 3

INTERVENTIONS:
Other: Observational Phase 1 — Noninterventional study
  Groups: Observational Phase 1
Other: Observational Phase 2, Group I — Noninterventional study
  Groups: Observational Phase 2, Group I
Other: Observational Phase 2, Group II — Noninterventional study
  Groups: Observational Phase 2, Group II
Other: Observational Phase 3 — Noninterventional study
  Groups: Observational Phase 3

SUMMARY:
This study gathers information for the development of a COPD care pathway for patients with cancer that reduces the treatment burden of patients, implements critical components of COPD care, and overcomes common barriers to COPD care in the community oncology clinic.

DETAILED DESCRIPTION:
Primary Objective: To design a feasible COPD care pathway for patients with cancer that reduces the treatment burden of patients, implements critical components of COPD care, and overcomes common barriers to COPD care in the community oncology clinic.

Secondary Objectives:

* To identify, characterize, and explain the treatment burdens of COPD and cancer as comorbidities, as reported by patients and providers.
* To identify, characterize, and explain barriers to COPD care in the oncology clinic, as reported by patients and providers.
* To identify, characterize, and explain important and feasible components of COPD care for patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* The participant has personal experience with medical management of COPD, defined as meeting at least one of the following criteria:

  1. patient with clinical documentation of COPD (either as a confirmed or suspected diagnosis) and has received at least one dose of an immune checkpoint inhibitor for cancer or
  2. provider who currently works at least part-time in a medical oncology clinic or
  3. provider who works at least part-time to care for patients with known or suspected COPD.

     A suspected diagnosis of COPD can be based on finding(s) by history, exam, or radiography (e.g., CT changes such as emphysema, bronchial wall thickening, or mucus plugging). A provider is defined as a physician, advanced practice provider, nurse, or respiratory therapist. Study team members are permitted to participate in the study if they meet eligibility criteria.
* Ability to understand and agree to participate on the study as described by the study information sheet.
* Capability of speaking or reading English.

Exclusion Criteria: Severe psychiatric symptoms; unusual social situation; or critical instability that would limit adherence to the study requirements, as determined by the study team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with clinical documentation of COPD and has received at least one dose of an immune checkpoint inhibitor for cancer or provider who currently works at least part-time in a medical oncology clinic or to care for patients with known or suspected COPD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Designing a Novel COPD Care Pathway | 12 months
  The feasibility of designing a novel COPD care pathway for patients with cancer that is responsive to mixed methods data by specifically addressing (i) the reduction of treatment burden of patients, (ii) the implementation of important and feasible components of COPD care, and (iii) the adaptation necessary to overcome common barriers to COPD care in the community oncology clinic, with feasibility defined by the agreement of a supermajority of stakeholders at a design team workshop.

SECONDARY OUTCOMES:
Number of Treatment Burdens Identified | 12 months
  Treatment burdens of COPD and cancer as comorbidities will be measured by self-report from patients and providers using surveys, interviews, and guided tours from at least one timepoint, with follow-up data collected from some participants.
  The options for the multiple-choice survey questions are based on historical data reporting the following specific features of COPD among patients without cancer: (i) inconsistent knowledge of the diagnosis of COPD,22 (ii) negative connotations of the diagnosis of COPD upon identity, (iii) lack of confidence in the capability of treating COPD, (iv) variable confidence in the skill of self-administering an inhaler, (v) inconsistent behavioral regulation for self-management of COPD, (vi) a goal to consolidate care to fewer appointments, (vii) lack of optimism for the ability to effectively treat COPD for positive consequences, and (viii) intention to utilize expanded access to COPD care.
Number of Barriers to COPD Care in Oncology Clinics | 12 months
  Barriers to COPD care in the oncology clinic will be measured by self-report from patients and providers using surveys, interviews, and guided tours from at least one timepoint, with follow-up data collected from some participants
  A quantitative analysis of barriers to COPD care using the data from multiple-choice survey answers of patients and providers to identify which types of barriers are most commonly experienced. The options for the multiple-choice survey questions are based on historical data reporting the following barriers to COPD care among patients without cancer: (i) inadequate information for providers or (ii) patients, (iii) lack of time, (iv) patients having a lack of faith in providers, (v) medical advice that conflicts with patients' perceptions, (vi) a desire for personal responsibility, and (vii) prohibitive cost of COPD care.
Identifying Important and Feasible Components of COPD Care - Best Practices for Cancer Patients | 12 months
  Important and feasible components of COPD care for implementation by a novel care pathway at community oncology clinics will be measured by qualitative and quantitative data collected from oncology patients and providers from at least one timepoint, with follow-up data collected from some participants. Participants will integrate this data using a concept mapping exercise to sort and rank items to identify COPD best practices among patients with cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lycan, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lycan TW Jr, Price SN, Mileham K, Stoen E, Ruiz J, Ohar JA, Norton D, Koch AL, Petty WJ, Birken SA. User-centered design of a COPD care pathway for patients with cancer: a mixed-methods clinical trial protocol. Future Oncol. 2025 Oct;21(25):3259-3273. doi: 10.1080/14796694.2025.2562715. Epub 2025 Oct 14. PMID 41084760